CLINICAL TRIAL: NCT06341530
Title: Prospective Clinical Study of Anlotinib Hydrochloride Capsule Combined With Penpulimab Injection in the Front-line Treatment of Advanced Non-small Cell Lung Cancer Patients
Brief Title: Anlotinib Combined With Penpulimab as Front-line Treatment in Advanced Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Chengzhe, Chief physician, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SURPASS-1
Record Dates: First submitted 2024-03-12; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — penpulimab; Immunotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Anlotinib combined with penpulimab
  Interventions: Drug: anlotinib combined with penpulimab

INTERVENTIONS:
Drug: anlotinib combined with penpulimab — single arm
  Other Names: Anti-angiogenesis combined with immunotherapy

SUMMARY:
In recent years, with the emergence and clinical application of anti-angiogenesis therapy, the therapeutic effect of patients has been significantly improved while ensuring that the adverse reactions of patients do not increase. Anti-angiogenic therapy can improve the hypoxia state of tumor tissue, normalize blood vessels, relieve immune suppression in tumor microenvironment, increase the degree of infiltration of immune cells, and fully activate immune cells to achieve the effect of tumor immunity. Previous studies have shown that penpulimab injection combined with anlotinib in the treatment of NSCLC can induce the normalization of tumor blood vessels and reshape the tumor immunosuppressive microenvironment, and the combination of the two can have synergistic effects.

This study intends to treat patients with advanced non-small cell lung cancer (NSCLC) confirmed by pathology with the combination of anlotinib and penpulimab injection, and observe the efficacy and safety of anlotinib and penpulimab injection in the first and second lines of NSCLC. This study is expected to provide a reference for the treatment strategy of advanced non-small cell lung cancer patients, and has important clinical value for the treatment of advanced lung cancer.

DETAILED DESCRIPTION:
This study intends to treat patients with advanced non-small cell lung cancer (NSCLC) confirmed by pathology with the combination of anlotinib and penpulimab injection, and observe the efficacy and safety of anlotinib and penpulimab injection in the first and second lines of NSCLC. To describe the therapeutic mode of anlotinib hydrochloride combined with penpulimab injection in the treatment of patients with non-small cell lung cancer (including treatment regimen, dosage, number of treatment cycles, dose adjustment/discontinuation and reasons) and treatment outcomes.Primary endpoints: Progression-free survival (PFS), disease control rate (DCR), objective response rate (ORR). Secondary endpoints: Overall survival (OS), quality of life score (QoL). Safety evaluation indicators: vital signs, laboratory indicators, adverse events (AE), serious adverse events (SAE).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old (calculated on the date of signing the informed consent);
* ECOG PS: 0-1;
* Expected survival ≥3 months;
* histopathologically confirmed non-small cell lung cancer with at least one measurable lesion (according to RECIST 1.1);
* Patients who provided detectable specimens (tissue or cancerous pleural fluid) for genotype testing before enrollment, and whose EGFR and ALK gene test results were negative; Or patients with negative test results; Or patients with positive test results and who are resistant or intolerant after receiving relevant targeted drug therapy.
* Have not been treated with a systematic regimen;
* Patients voluntarily join the project and sign informed consent;
* The function of vital organs is normal
* Physicians can benefit from anrotinib hydrochloride combined immunotherapy based on current clinical practice assessment;
* Patients voluntarily join the project and sign informed consent;
* Require initiation of antirotinib hydrochloride combined immunotherapy within 28 days of informed consent;

Exclusion Criteria:

* Known allergy or metabolic disorder to any drug in the treatment regimen;
* Those who refuse to take reliable contraceptive methods during pregnancy and lactation or in the appropriate age period;
* Have any history of uncontrolled medical diseases (including uncontrolled diabetes, severe heart, lung, liver and kidney dysfunction, blood, endocrine system diseases, and other malignant tumors);
* Have a history of psychotropic substance abuse, alcoholism or drug use;
* Currently or about to participate in other anti-tumor drug clinical trials;
* Have active, known, or suspected autoimmune diseases (including but not limited to: uveitis, enteritis, hepatitis, pituitaritis, nephritis, vasculitis, hyperthyroidism, hypothyroidism, and asthma requiring bronchodilator treatment, etc.). Patients with hypothyroidism who only need hormone replacement therapy, skin conditions that do not require systemic treatment (such as vitiligo, psoriasis, or alopecia) may be included;
* During the 6 months prior to entering the study, the following conditions occurred: Myocardial infarction, severe/unstable angina pectoris, NYHA grade 2 or higher cardiac dysfunction, poorly controlled arrhythmias (including QTcF interphase >450 ms in men, > 470 ms in women, >450 ms in women, >450 ms in men, > 470 ms in women, QTcF interval calculated by Fridericia formula), symptomatic congestive heart failure, cerebrovascular accident (including transient ischemic attack or symptomatic pulmonary embolism);
* Patients receiving hematopoietic stem cells or organ transplants;
* Other factors that may affect patient safety or compliance as determined by the investigator. Such as a serious illness (including mental illness) requiring co-treatment, serious laboratory abnormalities, or other family or social factors. Severe hepatic and renal insufficiency as judged by researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Quaque 3 week±7 Days
  From initiation of the investigational drug to first recording of disease progression (PD) Or the time between the date of death, depending on which occurs first. If no disease progression is observed, the cut-off date should be the date of the last tumor measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Zhe Cheng, Zhengzhou, Henan, China